CLINICAL TRIAL: NCT03953521
Title: Neuronavigated Theta Burst Stimulation in Depression
Brief Title: Neuronavigated TBS in Depression
Acronym: neuronaviTBS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Interim analysis indicated no statistical difference between treatment arms.
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Berthold Langguth, MD, Ph.D., Head of Center II and out-patient clinic of the Department of Psychiatry and Psychotherapy, University of Regensburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-1231-101
Record Dates: First submitted 2019-05-14; First posted 2019-05-16 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- navigated (Experimental): Positioning of the coil according to neuronavigation (Mylius et al., 2013, Definition of DLPFC and M1 according to anatomical landmarks for navigated brain stimulation: Inter-rater reliability, accuracy, and influence of gender and Age, NeuroImage 78, 224-232).
  Interventions: Device: intermittent Theta burst stimulation
- F3 (Active Comparator): Positioning of the coil according to EEG (electroencephalography) electrode Position F3 (marking this Position on a head cap).
  Interventions: Device: intermittent Theta burst stimulation

INTERVENTIONS:
Device: intermittent Theta burst stimulation — Stimulation of the left dorsolateral prefrontal Cortex with a specific repetitive transcranial magnetic Stimulation protocol (intermittent Theta burst Stimulation) according to Blumberger et al., 2018, Effectiveness of theta burst versus high-frequency repetitive transcranial magnetic stimulation in patients with depression (THREE-D): a randomised non-inferiority trial. Lancet. 2018 Apr 28;391(10131):1683-1692.

SUMMARY:
In this randomized controlled trial we will treat 80 patients with depression with intermittent theta burst stimulation in two parallel arms. Both arms are active interventions differing with respect to positioning of the treatment coil - one arm with neuronavigation and one arm with targeting according to EEG Position representing the left dorsolateral prefrontal cortex. Randomisation will be balanced for in- and out-patients and for the treatment arms.

DETAILED DESCRIPTION:
Intermittent Theta burst Stimulation (iTBS) is a specific type of repetitive transcranial magnetic Stimulation (rTMS). rTMS of the left prefrontal cortex was shown to be effective in the treatment of Depression. Recent studies showed that iTBS probably is as effective as rTMS.

One possibility to increase to efficacy of rTMS/iTBS is to use neuronavigation. With neuronavigation the coil Position can be targeted with an accuracy in the range of millimeters. Furthermore the Stimulation Position can be ensured during one single session and over the course of the daily Treatments.

The aim of the present study is to investigate the benefit of neuronavigation in the Treatment of Depression with iTBS by using two arms one with targeting the Stimulation site with neuronavigation and one by using the EEG Position F3 as target by using head caps for marking the position.

ELIGIBILITY:
Inclusion Criteria:

* unipolar or bipoloar depressive Episode according to ICD-10
* at least moderate Depression according to Hamilton Depression Rating Scale or ICD-10
* if applicable stable medication with psychoactive compounds for out-patients
* if applicable no or stable Treatment for Depression during the course of the Trial
* residence in Germany and mother tongue German
* written informed consent

Exclusion Criteria:

* Meeting the contraindications for transcranial magnetic Stimulation or magnetic resonance Imaging (electic devices or metal implants in the Body, e.g. cardiac pace maker, Insulin ppump)
* neurological disorders (e.g. cerebrovascular Events, neurodegenerative disorder, epilepsy, brain malformation, severe head Trauma)
* addictive disorder with consumption in the last two years
* regular intake of benzodiazepines
* participation in another study parallel to the Trial
* pregnancy or breastfeading period
* psychiatric confinement

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-05-27 (Actual)

PRIMARY OUTCOMES:
HAMD | 4 weeks
  Hamilton Depression Rating Scale

SECONDARY OUTCOMES:
HAMD | 16 weeks
  Hamilton Depression Rating Scale
MDI | 16 weeks
  Major Depression Inventory
PHQ-9 | 16 weeks
  9-question depression scale from the Patient Health Questionnaire
WHOQOL-BREF | 16 weeks
  WHO Quality of life scale (abbreviated Version)
CGI | 16 weeks
  Clincial Global Impression change

CONTACTS AND LOCATIONS:
Overall Officials: Berthold Langguth, PhD, Principal Investigator — University of Regensburg
Locations (1):
- Department of Psychiatry and Psychotherapy, University of Regensburg, Regensburg, Germany

REFERENCES:
- [Derived] Hebel T, Gollnitz A, Schoisswohl S, Weber FC, Abdelnaim M, Wetter TC, Rupprecht R, Langguth B, Schecklmann M. A direct comparison of neuronavigated and non-neuronavigated intermittent theta burst stimulation in the treatment of depression. Brain Stimul. 2021 Mar-Apr;14(2):335-343. doi: 10.1016/j.brs.2021.01.013. Epub 2021 Jan 22. PMID 33493624